CLINICAL TRIAL: NCT02320578
Title: Prospective Randomized Trial on2D Versus 3D Laparoscopic Radical Hysterectomy With Pelvic Lymphadenectomy for the Treatment of Early Stage Cervical Cancer (FIGO Stages IA2-IB1-IIA<2cm) and Advanced Stage Cervical Cancer (FIGO Stages IB2-IIA>2 Cm-IIB) Submitted to NACT With Complete Clinical Response.
Brief Title: 2D Versus 3D Radical Laparoscopic Hysterectomy for Cervical Cancer: a Prospective Randomized Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Catholic University of the Sacred Heart (Other)
Collaborators: Fanfani, Francesco, M.D. (Individual); Fagotti, Anna, M.D. (Individual)
Responsible Party: Principal Investigator, Prof. Giovanni Scambia, Director, Dip per la Tutela della Salute della Donna e della Vita Nascente, del Bambino e dell'Adolescente, Catholic University of the Sacred Heart
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 3D vs 2D Cervix
Record Dates: First submitted 2014-12-10; First posted 2014-12-19 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-06

CONDITIONS: Uterine Cervical Neoplasms; Laparoscopic Surgical Procedures
Keywords: Neoadjuvant Chemoptherapy; Laparoscopy 3D; Cervical cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 3D Laparoscopy (Experimental): Laparoscopic radical hysterectomy with pelvic lymphadenectomy are performed with 3D Laparoscopic technology.
  A 10 mm port is inserted at the umbilicus for the telescope. Once pneumoperitoneum (12 mmHg) is achieved, intra-abdominal visualization will be obtained with a 0° high-definition 3D telescope. Two additional 5 mm ports are placed under direct visualization. One more 5- mm trocar is inserted in the right mid abdomen at the level of the umbilicus. The instruments used include bipolar grasper, monopolar scissors, monopolar hook, various graspers and a suction irrigation system.
  Interventions: Procedure: 3D Laparoscopy
- Standard Laparoscopy (Active Comparator): Laparoscopic radical hysterectomy with pelvic lymphadenectomy are performed with standard laparoscopy technology. A 10 mm port is inserted at the umbilicus for the telescope. Once pneumoperitoneum (12 mmHg) is achieved, intra-abdominal visualization will be obtained with a 0° high-definition telescope. Two additional 5 mm ports are placed under direct visualization. One more 5 mm trocar is inserted in the right mid abdomen at the level of the umbilicus. The instruments used include bipolar grasper, monopolar scissors, monopolar hook, various graspers and a suction irrigation system.
  Interventions: Procedure: Standard Laparoscopy

INTERVENTIONS:
Procedure: 3D Laparoscopy — 3D Laparoscopy approach
  Arms: 3D Laparoscopy
Procedure: Standard Laparoscopy — Standard laparoscopy approach
  Arms: Standard Laparoscopy

SUMMARY:
The aim of this prospective randomized pilot study is to verify if the operative time of a Radical abdominal hysterectomy (LRH) with pelvic lymphadenectomy for early stage cervical cancer (FIGO stages IA2-IB1-IIA<2cm) and for advanced stage cervical cancer (FIGO stages IB2-IIA>2cm-IIB) submitted to neoadjuvant chemotherapy (NACT) with complete clinical response could be further reduced using 3D Laparoscopy (Olympus Medical Systems Corp) versus standard laparoscopy

DETAILED DESCRIPTION:
Radical abdominal hysterectomy (RAH) with pelvic lymphadenectomy is the standard surgical treatment for early stage cervical carcinoma FIGO stages IA2-IB1-IIA<2cm. Since the early 90's laparoscopic radical hysterectomy with pelvic lymphadenectomy (LRH) has been suggested as surgical approach for the treatment of cervical cancer. In the recent years, many institutions have begun to consider it an attractive technique and to study its feasibility and safety. Most of these studies have shown that LRH is relatively more time-consuming than standard laparotomy and ranges from 90 to 420 minutes according to surgeons' experience and different techniques adopted to achieve hemostasis, resect the parametrium and uterosacrals. Spirtos et al. demonstrated that staplers could reduce mean operation time from 253 to 205 minutes if compared to argon beam coagulator. Moreover, the pulsed bipolar system was associated with significant reduction in operative time in comparison with the conventional bipolar system (mean, 172 minutes vs 229 minutes; P < 0.001). The largest series of LRH reported from a single institution by Puntambekar et al included 248 patients and described the "Pune technique" (anterior and posterior peritoneal U cuts, early dissection of the rectovaginal space, fully mobilization of the uterus, resection of the cardinal and uterosacral ligaments with Ligasure system (Ligasure Vessel Sealing System; Valleylab, Tyco Healthcare, Boulder, CO)), obtaining a very short mean operative time (mean, 92 minutes; range 6-120 minutes).

A recent review on laparoscopic and robot-assisted radical hysterectomy with pelvic lymphadenectomy including 17 studies reported a mean operating time of 202 minutes [range, 184-221 minutes] in the group of LRH, which matches with our experience of 210 min (range 180-240), using conventional bipolar electrosurgery.

This prospective randomized pilot study is aimed to verify if the operative time of a LRH with pelvic lymphadenectomy for early stage cervical cancer (FIGO stages IA2-IB1-IIA<2cm) and for advanced stage cervical cancer (FIGO stages IB2-IIA>2cm-IIB) submitted to neoadjuvant chemotherapy (NACT) with complete clinical response could be further reduced using 3D Laparoscopy (Olympus Medical Systems Corp) vs. standard laparoscopy.

Saving operative time would mean shorter anesthesia and faster recovery, further improving the safety profile of the laparoscopic approach in the treatment of cervical cancer.

Secondary endopoints of this comparison are incidence of intra- or postoperative complications (Cardiac, Respiratory, Neurological, Gastrointestinal, Renal, Fever, Wound or other Infection, Lymphocele), estimated blood loss, days of hospitalization and costs for the health care system.

ELIGIBILITY:
* Age ≤ 75 years
* Patient's informed consent
* American Society of Anesthesiologists: < class III or IV
* No actual pregnancies or P.I.D.
* No previous major abdominal surgical procedures
* Early stage cervical cancer (FIGO stages IA2-IB1-IIA<2cm) and advanced stage cervical cancer (FIGO stages IB2-IIA>2cm-IIB) submitted to NACT with complete clinical response
* No previous radiotherapy on the pelvic field
* No uterine size larger than conform 10 weeks gestation

Max Age: 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2014-10; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Operative time for laparoscopic radical hysterectomy with pelvic lymphadenectomy | Intraoperative
  Operative time will be calculated from the entrance in the abdominal cavity to the closure of the skin trocar accesses

SECONDARY OUTCOMES:
Number of participants with intra or post operative complications | two years
  Cardiac, Respiratory, Neurological, Gastrointestinal, Renal, Fever, Wound or other Infection, Lymphocele

CONTACTS AND LOCATIONS:
Locations (1):
- Catholic University of the Sacred Heart, Rome, Italy, Italy